

#### INFORMED CONSENT TO TAKE PART IN A RESEARCH STUDY

**TITLE OF STUDY:** Immediate Versus Delayed Insertion of Nexplanon after

Termination of Pregnancy Over 14 Weeks Gestation (The

NAPA Study)

#### **INVESTIGATORS:**

PRINCIPAL INVESTIGATOR: Allison A. Cowett, MD, MPH

Associate Medical Director Family Planning Associates Medical Group

659 West Washington Boulevard

Chicago, IL 60661

Telephone: 312-707-8988

#### SUB-INVESTIGATORS:

Rose Ali, PA-C

First Clinician

Family Planning Associates Medical Group

#### Mark Evans, MSPH

University of Pittsburgh School of Medicine 3550 Terrace Street Pittsburgh, PA 15261

Telephone: 412-648-9040

#### PHYSICIAN CONSULTANT

Miriam Cremer, MD, MPH

Staff physician, Cleveland Clinic Director of Global Health Research,

Obstetrics, Gynecology & Women's Health Institute

Telephone: 412-641-5496

PHONE NUMBER: 312-707-8988

SPONSOR: Merck & Co., Inc.

#### What is the purpose of this form?

You are being asked to participate in a research study. It is important that you read the following explanation of the proposed procedures. This form describes the purpose, procedures, benefits, risks, discomforts, and precautions of the study. It also describes the alternative procedures that are available to you and your right to withdraw from the study at any time. A member of the study staff will read through the consent with you and discuss all the information. When you think you understand the study, you will then be asked if you agree to take part. If you agree, you will be asked to sign this consent form. Once you sign it, we will give you a signed and dated copy to keep.

#### Why is this study being done?

Nexplanon is an FDA-approved form of reversible birth control (meaning that your chance of getting pregnant after it is discontinued or removed is similar to women not using birth control). Usually, Nexplanon is placed 3 to 4 weeks after a second trimester surgical abortion. However, we think that it is possible that there will be a higher rate of continued use of Nexplanon six months after the second trimester surgical abortion if it is placed immediately after that procedure.

#### What is being studied?

This study is testing the timing of Nexplanon placement after a second trimester surgical abortion.

You are being asked to be in this study because you have chosen to have a second trimester surgical abortion and you have indicated that you would like to use Nexplanon for contraception afterward.

The device being studied is approved by the FDA for pregnancy prevention. Once your participation in the study is complete, you will be able to continue to use the Nexplanon for up to three (3) years after the device was inserted.

# Who is being asked to take part in this research study?

You are being asked to take part in this study because you are a woman 18 years of age and older, are between 14 0/7 and 23 6/7 weeks pregnant, are scheduled to have a second trimester surgical abortion, desire a Nexplanon for contraception, and have no medical problems that would prevent you from receiving Nexplanon. About 120 women will be participating in this study. As the standard practice is to place Nexplanon 3 to 4 weeks after a second trimester surgical abortion, you will be asked by your care provider to choose another form of birth control to use during that time. Your care provider will have discussed all methods of birth control that you can use. The method of birth control that you

choose may be a non-hormonal form of birth control such as abstinence (not having sex), condoms, or spermicide or you may request a hormonal method of birth control, such as the birth control pill.

If you are randomly (by chance) assigned to receive your Nexplanon immediately after the second trimester surgical abortion, you will not need to use this other form of birth control. If you are randomly (by chance) assigned to receive your Nexplanon 2 to 4 weeks after the second trimester surgical abortion, you will need to use this form of birth control until that visit.

#### What do I need to know about this study?

About 120 subjects will take part in this study, which will only be conducted at this location. The entire study will last for about 1 year. Your participation in the study will be about 6 months.

#### What will happen during this study?

During this study, you will have:

- From 1 to 3 office visits
- Each office visit will be up to 4 weeks apart
- This study will have 2 different groups one group will receive Nexplanon right after their second trimester surgical abortion and the other group will receive it at a follow-up visit. This other group will be provided with another method of birth control to use until the follow-up visit.
- You will be randomly (by chance) assigned to a study group by a process similar to flipping a coin. You have an equal chance (a 50/50 chance) of being in either group.

### **Details of Procedures:**

If you decide to take part in this research study, you will undergo the procedures listed below. If you decline to participate, de-identified data (data that cannot be linked to you) will be maintained regarding why you declined.

# **Screening/Enrollment Procedures**

Procedures to determine if you are able to take part in a research study are called "screening procedures". For this research study, the screening procedures will take place in the FPA clinic where you see your care provider and will take about 1 hour.

Before any study-related tests and procedures are performed, you will be asked to read and sign this consent form, which is for all study procedures.

#### <u>Screening Procedures:</u>

- 1. A research clinician will review all of your birth control options again and confirm that you plan to use Nexplanon for birth control after your second trimester surgical abortion.
- 2. A research clinician will also ask you some information about your background general health and pregnancy history, birth control history, as well as your current use of any medications.
- 3. A research staff member will ask you some questions about health insurance.
- 4. A research staff member will give you a form with some questions about partner violence and forced sex or forced pregnancy for you to fill out in private.
- 5. A research clinician will take your blood pressure, height, and weight.
- 6. Results of your general appearance and other body systems will be noted, as well as any contraceptive counseling you receive.

### **Experimental Procedures:**

If you qualify to take part in this research study, you will undergo the experimental procedures, listed below, on the day of your second trimester surgical abortion.

- When your second trimester surgical abortion is completed, your doctor will check that you did not have any medical complication related to the procedure, and are okay to have the Nexplanon placed. If you are not okay to have the Nexplanon placed after the second trimester surgical abortion is complete, you will no longer be able to participate in the research study. Arrangements will be made by your physician for follow-up care as necessary. You can use an alternate form of birth control until that time.
- If the doctor can place the Nexplanon the doctor will open an envelope assigned to you at random (by chance) to see if you are to get the Nexplanon immediately after your second trimester surgical abortion or you are to come

back in 2-4 weeks to have the Nexplanon placed. The process of being placed in one of these two groups is like flipping a coin. You have a 50/50 chance of being assigned into either of the two groups. You will not find out which group you have been assigned to until you have completed your second trimester surgical abortion.

- If you are assigned into the group who has their Nexplanon placed at the time of the second trimester surgical abortion (Group 1), the doctor will place your Nexplanon immediately after your procedure, before you wake up, in a standardized manner.
- o If you are assigned to the group who has the Nexplanon placed at your follow up visit (Group 2), you will be given a follow up appointment on the day of your procedure to return to the Family Planning Associates office in 2 to 4 weeks after your second trimester surgical abortion to have your Nexplanon placed. The visit will take approximately 2 hours to complete. You will use the alternate form of birth control you discussed with the clinician until you return for your insertion visit.
  - You will receive one reminder phone call, text message or email from the Research Office staff prior to this visit.
  - During this visit, you will have your Nexplanon placed. Your blood pressure, height, and weight will be taken. You will be asked some questions about your return for the Nexplanon implant. If needed, a small amount of urine will be collected in order to have a pregnancy test.

# Procedure for insertion of the implant:

If you are receiving your Nexplanon immediately after the abortion, you will be asleep for the insertion. If you are selected to receive your Nexplanon at a follow-up visit, a numbing agent will be used prior to the insertion of the implant. After numbing the area, an applicator will be inserted into your arm and a purple slider will be pulled back to release the implant into your arm. Information related to the Nexplanon insertion will be placed into your medical record. Some of the information from your medical record may be obtained for the research record. None of the research record will be placed into your medical record chart.

# Monitoring/Follow-up Procedures:

Procedures performed to evaluate the effectiveness and safety of the experimental procedures are called "monitoring" or "follow-up" procedures. For this research study both groups will take part in a follow-up phone call. The monitoring/follow-up procedures include:

1. Six months after the second trimester surgical abortion, we will contact you in order to complete a telephone survey. This will include questions about your current medical history, your experience with the Nexplanon, and how you are currently feeling. You will be asked to feel for the implant in your arm while on the phone. In the rare case that you cannot feel the implant, you will be brought in for a clinical evaluation. You will be contacted at this time regardless of whether you have returned for any of your other follow-up appointments. If you still desire Nexplanon for contraception, you will be referred to either a hospital clinic or your private doctor for the Nexplanon placement.

At any time during this study, you will be able to contact the Family Planning Associates office with questions or to make an unscheduled visit. If you have any complaints, concerns of infection, or suspect pregnancy, you can call and schedule an appointment to follow up.

# What are the potential risks, side effects, and discomforts of being in the study?

There may be some possible risks and discomforts from being part of this study.

- 1. *Emotional Discomfort*: Some of the questions you will be asked may make you feel uncomfortable or upset. You may refuse to answer any question at any time. Counseling referrals are available if you need help at any time.
- Participating in research: Participation in a research study may be inconvenient or cause a breach of confidentiality, meaning that others may find out you are participating in this study. Research staff will do everything possible to protect your privacy.
- 3. Risk with Nexplanon insertion and removal: The implant may not be placed in your arm due to a failed insertion. If this happens, you may become pregnant. If you think you are pregnant, you should see your health care provider and contact the study team as soon as possible. Continuing to have the Nexplanon implanted while pregnant may be dangerous. The physician who inserts your Nexplanon will feel your arm immediately after placement to be sure that it is possible to feel the implant. When you remove the bandage the day following your surgery you should be able to feel the implant. If you cannot feel the implant you should contact the clinician immediately.

Every effort will be made to correctly insert your implant. Removal of the implant may be difficult or impossible if it is not placed where it should be. Special procedures, including x-rays, CT scans, MRIs, blood tests or surgery, may be needed to detect and/or remove the implant if it is not placed in the proper location.

#### Other risks with insertion and removal are as follows:

- Pain, irritation, swelling, or bruising at the insertion site.
- Scarring, including a thick scar called a keloid may appear around the insertion site. Scar tissue around the insertion site may make it more difficult to remove the implant.
- Risk of infection at the insertion site.
- Risk of discomfort during insertion.
- The need for surgery to remove the implant.
- Risk of injury to the nerves or blood vessels in your arm where the implant is placed.
- The implant may break making the removal difficult.
- Risk of local anesthesia: there is an uncommon risk of getting an unusual taste in your mouth, ringing in your ears, nausea or lightheadedness from the numbing medicine used in your arm for the insertion and removal. Rarely, you can have a seizure or death from the numbing medicine.

# 4. Side effects and risks with Nexplanon use:

- The most common side effect is a change in the menstrual cycle. Many women will experience irregular bleeding after Nexplanon insertion. Other changes include: mood swings, weight gain, headaches, acne, and depressed mood.
- Other side effects include: breast pain, amenorrhea (absence of periods), nervousness, back pain, nausea, dizziness, pain, and pain at the insertion site.
- Failure to prevent pregnancy is a rare risk. If you think you are pregnant, you should see your health care provider as soon as possible.

As with any experimental procedure, there may be adverse events or side effects that are currently unknown and could be permanent, severe, or life threatening. A research doctor is available 24 hours a day; every day of the week, at 312-707-8988 in case you have any questions or need to report any problems. You will

be informed of any new and significant side effects, or any other information that may affect your willingness to continue in the study.

#### Will you be informed of new information relating to the study?

All new findings discovered during the course of this research study that may reasonably affect your health and welfare and/or might change your decision to continue to participate in this study will be provided to you by your study doctor as such information becomes available. You may be asked to sign a new consent form to continue in the study if this happens.

#### Does being in this study provide any benefit?

This research study is designed to select by chance the timing of receiving birth control. You may or may not benefit from your participation in this study.

### Whom do you contact in the event of an emergency?

If you experience an adverse reaction or a research-related injury during the course of the study, you should immediately contact Dr. Cowett of FPA at 312-707-8988.

If you seek emergency care, or if you are hospitalized, please alert the doctor who is treating you that you are enrolled in this research study being conducted by Dr. Cowett of Family Planning Associates.

# What happens if you have a research related injury?

If you believe that you are injured as a result of the research procedures being performed, please contact the Principal Investigator or one of the co-investigators listed on the first page of this form immediately. You may receive medical care in the same way as you would normally. Emergency medical treatment for injuries solely and directly related to your participation in this research study will be provided to you by the hospitals to which Family Planning Associates refers patients. It is possible that a hospital may bill your insurance provider for the costs of this emergency treatment, but none of these costs will be charged directly to you. If your research-related injury requires medical care beyond this emergency treatment, you will be responsible for the costs of this follow-up care unless otherwise specifically stated below. There is no plan for monetary compensation (such as for lost wages, lost time, or discomfort). You will not, however, be giving up any of your legal rights by signing this consent form.

# What other treatments or procedures are available if you decide not to take part in this research study?

You can refuse to be in this research study. If you refuse to be in this study, you will still be able to receive any of the services otherwise available to you at Family Planning Associates or through your own doctor. Your second trimester surgical abortion will be done in the usual manner and you will have the option of using other forms of birth control currently offered by Family Planning Associates outside of the research study.

#### Will it cost you anything to be in this study?

You will be receiving medical care as a part of this research study. Nexplanon implant and insertion will be provided at no cost to you as part of participation in the study. The study-related activities and study visits will be provided at no charge to you or your insurance company while in the study. If you receive a bill or believe that your health insurance has been billed for something that is part of the research study, notify a member of the research team or any Family Planning Associates staff member. You and/or your health insurance will be charged in the standard manner for services and procedures provided for your routine care, including your second trimester surgical abortion. If surgery is needed to remove the Nexplanon, the study will pay for the procedure. You will need to pay any costs for medical care for problems not related to the use of the study product. You will need to pay any costs for any visits to the Emergency Room not authorized by one of the researchers unless immediate medical care is needed. The phone call at 6 months is for research only and neither you nor your insurance will be charged for this. If you choose to continue using Nexplanon after the study ends, you will be responsible for any costs associated with the implant.

# Will you be paid for being in this study?

You will be reimbursed for taking part in the study. The money will pay for your inconvenience and time off work.

You will be reimbursed a total of \$100 (Group 1) or \$115 (Group 2) if you complete all parts of this study. The terms of this reimbursement are:

- \$75 for completing the screening/enrollment visit, including all of the study procedures
- \$15 for completing the follow-up visit to get Nexplanon (Group 2, delayed group only)
- \$25 for completing the 6-month telephone follow-up. As long as you complete the 6-month telephone call you will receive the \$25 payment. If

you are in Group 2 and you do not return for your Nexplanon, you can still receive payment if you complete the follow-up phone call.

If you complete part, but not all of the study, you will receive partial payment based on the visit that you have completed as outlined above. A complete visit or phone call requires that all study procedures get done and all questionnaires are completed. Partial visits will not be reimbursed.

Reimbursements made to you for taking part in this study will be reported to the IRS as income as required by law, so you are required to provide your social security number. No deductions for any state or federal withholding or any other similar taxes will be made. It is your responsibility to report this compensation on state and federal tax returns and for the payment of any taxes that are due on this compensation.

#### Do you have to be in this study?

Your participation in this research study, to include the use and disclosure of your identifiable information for the purposes described above, is completely voluntary. (Note, however, that if you do not provide your consent for the use and disclosure of your identifiable information for the purposes described above, you will not be allowed to participate in the research study.) Whether or not you provide your consent for participation in this research study will have no effect on your current or future relationship with Family Planning Associates. Whether or not you provide your consent for participation in this research study will have no effect on your current or future medical care at Family Planning Associates or on your current or future relationship with a health care insurance provider.

Your doctor may be involved as an investigator in this research study. As both your doctor and a research investigator, s/he is interested both in your medical care and the conduct of this research study. Before agreeing to participate in this research study, or at any time during your study participation, you may discuss your care with another doctor who is not associated with this research study. You are not under any obligation to participate in any research study offered by your doctor. You also have the right to request that your questions, concerns, or complaints be addressed by a physician investigator involved in this research.

Your refusal to participate or your withdrawal from the study will involve no penalty or loss of benefits to which you are entitled. You may stop your participation at any time without affecting your ongoing medical care.

# Can you withdraw, at a future date, your consent for participation in this research study?

You may withdraw, at any time, your consent for participation in this research study, to include the use and disclosure of your identifiable information for the purposes described above. (Note, however, that if you withdraw your consent for the use and disclosure of your identifiable medical record information for the purposes described above, you will also be withdrawn, in general, from further participation in this research study.) Any identifiable research or medical information recorded for, or resulting from, your participation in this research study prior to the date that you formally withdrew your consent may continue to be used and disclosed by the investigators for the purposes described above.

You can always withdraw your authorization to allow the research team to review your medical records by contacting the investigator listed on the first page, and making the request in writing.

Your decision to withdraw your consent for participation in this research study will have no effect on your current or future relationship with Family Planning Associates. Your decision to withdraw your consent for participation in this research study will have no effect on your current or future medical care at Family Planning Associates or your current or future relationship with a health care insurance provider. If you choose to withdraw from the study, you will have to follow up with your physician in order to continue to get birth control.

# Can you be removed from the study without your permission?

If you agree to take part in this research study, an Investigator can ask you to stop participating in the study without your permission for the following reasons:

- 1) You decide to not terminate the pregnancy.
- 2) You show up for the 'delayed' insertion visit outside of the 2-4 week window, and have a positive pregnancy test.
- 3) You do not follow all of the study instructions.
- 4) The researchers feel it is in your best interest because of a personal or medical condition.
- 5) You have a serious reaction or health problem related to being in the study.
- 6) Study enrollment is stopped or the study is canceled.

We will continue to use any research or medical information that was obtained prior to your removal from the study. There is no risk to you from stopping the study early.

# As part of this study, we are also requesting your authorization or permission to review your medical records to obtain past and current medical information from Family Planning Associates' records.

We will obtain information concerning your diagnosis, age, past medical history, diagnostic procedures, and results of any blood tests that were already done as part of your standard medical evaluations at Family Planning Associates clinics. We will use this information to determine whether you meet the conditions for participation in this study, to compare your earlier test results to the findings from this study and, if necessary, to use your previous exam results in place of or in addition to some of the exams needed for this study. The results of any visits that you make to the Emergency Department at an outside hospital because of issues related to the study will become part of your medical records at the hospital. All other information gathered during this study will only be kept in the Family Planning Associates office as described above.

#### Who will have access to your study and/or medical information?

Any information about you obtained from this research will be kept as confidential as possible. All records related to your involvement in this research study will be stored in a locked file cabinet in the Family Planning Associates office. Your records will be kept in such a way that it is possible to link the research data to your identity. Only the investigators and their research staff have access to the research records. However, the study doctor, the sponsor or it's designee and, under certain circumstances, the Food and Drug Administration (FDA) and New England Independent Review Board (IRB) will be able to inspect and have access to confidential data that identifies you by name. Information from the records will be entered into a computer database. For the computer records, your identity will be indicated by a participant identification number rather than by your name, and the information linking this number with your identity will be kept separate from the computer records. You will not be identified by name in any publication of the research results unless you sign a separate consent form giving your permission (release). By signing this consent form, you authorize the study doctor to release your medical records to the sponsor, the FDA, and the IRB.

In addition to the investigators listed on the first page of this authorization (consent) form and their research staff, the following individuals will or may have access to identifiable information (which may include your identifiable medical information) related to your participation in this research study:

- Authorized representatives of the New England IRB may review your identifiable research information (which may include your identifiable medical information) for the purpose of monitoring the appropriate conduct of this research study.
- In unusual cases, the investigators may be required to release identifiable information (which may include your identifiable medical information) related to your participation in this research study in response to an order from a court of law. If the investigators learn that you or someone with whom you are involved is in serious danger or potential harm, they will need to inform, as required by Illinois law, the appropriate agencies.
- Authorized representatives of the sponsor of this study, Merck, may review and/or obtain identifiable information (which may include your identifiable medical information) related to your participation in this research study for the purpose of monitoring the accuracy and completeness of the research data and for performing required scientific analyses of the research data. While the study sponsor understands the importance of maintaining the confidentiality of your identifiable research and medical information, Family Planning Associates and the Cleveland Clinic cannot guarantee the confidentiality of this information after it has been obtained by the study sponsor. The investigators involved in the conduct of this research study may receive funding from the sponsor to perform the research procedures and to provide the sponsor with identifiable research and medical information related to your participation in the study
- Authorized representatives of the U.S. Food and Drug Administration or the Office for Human Research Protections (OHRP) may review and/or obtain identifiable information (which may include your identifiable medical information) related to your participation in this research study for the purpose of monitoring the accuracy of the research data and to ensure the protection of research subjects. While the U.S. Food and Drug Administration and the OHRP understand the importance of maintaining the confidentiality of your identifiable research and medical information, Family Planning Associates and the Cleveland Clinic cannot guarantee the confidentiality of this information after it has been obtained by the U.S. Food and Drug Administration or the OHRP.
- Authorized representatives of Family Planning Associates may have access to identifiable information (which may include your identifiable medical information) related to your participation in this research study for the purpose of (1) fulfilling orders made by the investigators for hospital and

health care services (e.g., laboratory tests, diagnostic procedures) associated with research study participation; (2) addressing correct payment for tests and procedures ordered by the investigators; and/or (3) for internal clinic operations (i.e. quality assurance).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Will this research study involve the use or disclosure of your identifiable medical information?

The results of any separate visits that you make to an emergency room or doctor's office because of issues related to the study will become part of your medical records. All information gathered during this study will be kept only in the Family Planning Associates office as described above.

For how long will the investigators be permitted to use and disclose identifiable information related to your participation in this research study? The investigators may continue to use and disclose, for the purposes described above, identifiable information (which may include your identifiable medical information) related to your participation in this research study for a minimum of 7 years and for as long (indefinite) as it may take to complete this research study.

# Can you have access to your medical information that results from your participation in this research study?

In accordance with the Family Planning Associates' Notice of Privacy Practices document that you have been provided, you are permitted access to information (including information resulting from your participation in this research study) contained within your medical records filed with your health care provider.

# Whom do you contact if you have questions about the study? If you have questions or concerns about the study, you can contact Dr. Cowett at 312-707-8988.

If you have questions about your rights as a research subject, or other concerns about the research, you can contact NEIRB at 1-800-232-9570.

#### **VOLUNTEER'S STATEMENT:**

I agree that I have been given a chance to ask questions about this research study. These questions have been answered to my satisfaction. I may contact Dr. Cowett if I have any more questions about taking part in this study. Dr. Cowett or the company she is employed by is being paid by the sponsor for my participation in this study.

My participation in this research project is voluntary. I may quit the study at any time without harming my future medical care or losing any benefits to which I might be entitled. The investigator in charge of this study may decide at any time that I should no longer participate in this study.

If I have questions about my rights as a research subject, other concerns about the research, or I am unable to reach the investigator, I can contact:

New England IRB Telephone: 1-800-232-9570

By signing this form, I have not waived any of my legal rights.

I agree to participate in this study. I will be given a copy of this signed and dated form for my own records.

| Study Participant (signature) | Date |
|---------------------------------------------|----------|
| Print Participant's Name | |
| Person who explained this study (signature) | <br>Date |